CLINICAL TRIAL: NCT03010410
Title: Platelet Immune Responses in Aging and Influenza and Sepsis (INVACS)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Samuel Brown, Director, Center for Humanizing Critical Care, Intermountain Health Care, Inc.
Other Study IDs: 1040298
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Sepsis; Influenza
MeSH Terms: conditions — Sepsis; Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study will bank remaining platelet lysates for future assays.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Influenza/respiratory virus pts <65 yrs: Patients with a primary microbiologic diagnosis of influenza (any strain) or other routinely clinically identified respiratory viruses
- Influenza/respiratory virus pts ≥ 65 yrs: Patients with a primary microbiologic diagnosis of influenza (any strain) or other routinely clinically identified respiratory viruses
- Sepsis/septic shock patients < 65 yrs: Sepsis and septic shock patients
- Sepsis/septic shock patients ≥ 65 yrs: sepsis and septic shock patients

SUMMARY:
Aging is associated with immunosenescence and impaired host defense mechanisms, contributing to influenza-related morbidity and mortality. Preliminary data demonstrate that the platelet transcriptome is markedly different between healthy subjects and influenza patients. Interferon-induced transmembrane proteins (IFITM) family members are among the transcripts significantly increased in platelets during influenza and expression of IFITM-3 is impaired in elderly subjects, a pattern associated with increased mortality. This study will build on these data and investigate if aging influences the expression of platelet IFITM family members in patients with influenza and sepsis.

This study will prospectively determine if aging alters the induction of (IFITMs) in platelets from hospitalized influenza and sepsis patients. The study will also determine if diminished expression of IFITM family members correlates with an increased risk of adverse outcomes in older influenza and sepsis patients.

DETAILED DESCRIPTION:
This will be a prospective observational cohort study comparing older (age≥65) and younger (age<65) influenza and sepsis patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old at the time of enrollment
* Meet one of the following three main criteria:

A. INFLUENZA (AND OTHER RESPIRATORY VIRUS) PATIENTS:

Patients admitted to the intensive care unit (ICU) with a primary microbiologic diagnosis of influenza (any strain) or other routinely clinically identified respiratory viruses within 1 week of symptom onset. Influenza or other respiratory virus will be diagnosed using an RT-PCR viral panel on a respiratory tract specimen, as is currently standard of care on patients admitted to the ICUs at IMC with respiratory symptoms.

OR

B. SEPSIS PATIENTS:

Sepsis patients must have

1. Suspected or confirmed infection

   AND
2. Organ dysfunction as defined by a SOFA >= 2 above baseline (if no baseline data available, SOFA assumed to be 0)

OR

C. SEPTIC SHOCK PATIENTS:

AFTER INFUSION OF 20ML/KG CRYSTALLOID OR EQUIVALENT, Septic shock patients must have

1. Suspected or confirmed infection

   AND
2. Lactate > 2 mmol/L

   AND
3. Receiving vasopressors

   * All patients must be enrolled into the study within 72 hours of ICU admission

Exclusion criteria

* Have a congenital or acquired immunodeficiency disorder (e.g., chronic variable immune deficiency, agammaglobulinemia, hypogammaglobulinemia, leukocyte adhesion defects, IgA deficiency, etc.)
* Have neutropenia (<1,000/mm3)
* Have received immunosuppressant medications within the previous 30 days (e.g., prednisone or prednisone equivalent at a dose≥10mg daily for ≥14 days or any cyclosporine, TNF-alpha antagonists, tacrolimus, sirolimus, interferons, mycophenolate, biological agents, methotrexate, azathioprine, polyclonal/monoclonal antibodies, etc.)
* Have any history of bone marrow or organ transplantation
* Have an active malignancy (not including non-melanoma skin cancer or localized prostate cancer), or have received chemotherapy drugs within the last 6 months.
* Have been admitted to the ICU for greater than 72 hours
* Have a Hemoglobin level <7gm/dl
* Have clinically significant bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a prospective observational cohort study comparing older (age≥65) and younger (age<65) influenza and sepsis patients.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-12-21 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
90 day mortality | 90 days
  For the increased risk of mortality outcome, 90-day mortality will be the primary outcome variable. This will be modeled using mixed effects logistic regression, using days 0, 3, and 7 as repeated measurements. In this fashion, IFITM-3 and mortality are time-varying. A separate model will be fitted for the younger and older groups, since age group is expected to be collinear with IFITM-3 protein.

SECONDARY OUTCOMES:
28 day mortality | 28 days
  The same sample of influenza patients will be used for mortality analysis. Based on published and unpublished data, 28-day mortality in critically-ill influenza patients admitted to ICUs ranges from 10-40%, even during non-pandemic periods. Based on these estimates, our sample size (n=75 younger and n=75 older) provides 84% power (two-sided alpha 0.05 comparison) to detect a difference in incidence of 29% and 9%, which is a conservative estimate of the difference between the younger and older groups.
Interferon-induced transmembrane protein expression in platelets | 24(±12) hours of diagnosis (day 0 or 1), day 3, 5, and 90
  Recent evidence also demonstrates that IFITM-3 acts as a membrane organizer by facilitating clathrin-mediated endocytosis (CME). This membrane-organizing process allows cells to internalize molecules and viruses. CME regulates platelet membrane organization. IFITM-3 is demonstrated as necessary for host defenses against influenza virus. Moreover, with absent or reduced levels of IFITM-3, cells do not effectively restrict viral replication, an impaired response that may influence adverse clinical outcomes.
IFITM-3 mRNA | 24(±12) hours of diagnosis (day 0 or 1), day 3, 5, and 90.
  Platelet IFITM-3 protein levels have been seen to be increased in influenza patients and correlated with IFITM-3 mRNA (r2=0.33, p<0.005). However, in hospitalized influenza patients, platelet IFITM-3 mRNA and protein expression was decreased in older, compared to young patients.
  It is hypothesized that influenza will induce expression of IFITM family members in platelets; IFITM's expression will be reduced in older compared to young influenza patients. This hypothesis will be tested to determine whether or not influenza induces IFITM-3 expression in human platelets and compare older and young subjects. Here, an outcome of IFITM-3 protein will be tracked in conjunction with mRNA.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel M Brown, MD MS, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No